CLINICAL TRIAL: NCT04064385
Title: Functional Electrical Stimulation Cycling in Acute Spinal Cord Injury; a Feasibility Study
Brief Title: Functional Electrical Stimulation Cycling in SCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glasgow Caledonian University (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Aleksandra Dybus, REsearch Physiotherapist, Glasgow Caledonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GN19NE123
Record Dates: First submitted 2019-07-04; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Spinal Cord Injury, Acute; Paraplegia; Tetraplegia
Keywords: Functional Electrical Stimulation Cycling; Physical Therapy
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): FES cycle training will be performed on the RT300 FES cycle ideally 3 times per week for 6 weeks, each session lasting up to 90 minutes. Electrical stimulation will be delivered through up to 12 independent channels each delivering up to 140 mA current on the following muscles (both on the right and left leg): quadriceps, femoral biceps and gluteus, gastrocnemius and tibialis anterior. Abdominal and back extensor muscles may also be stimulated if the participant presents with neurological trunk weakness (SCI above T6). The FES unit will stimulate the muscles that extend the hip (gluteals), flex the knee (hamstrings) and extend the knee (quadriceps) in the correct order to bring about a cycling motion. The feet and lower legs of the participants will be strapped into the pedals and the wheelchair will be coupled in a rigid manner with the training device.
  Interventions: Device: FES Cycling
- Control (No Intervention): Participants in the control group will receive usual care, consistent with standard NHS care in this population. Usual physiotherapy care is provided, up to 2 times per day, 4 to 5 days per week, each lasting approximately 90 minutes. Physiotherapists provide one to one function-oriented physiotherapy session to improve balance, muscle strength and transfer skills.

INTERVENTIONS:
Device: FES Cycling — Stimulation parameters will be 450μs, 40Hz, and up to 140mA, these values will be changed if needed based on individual response. For example, stimulation to the gluteal muscles often may to be decreased to prevent autonomic dysreflexia. To receive correct stimulation parameters, stimulation intensity will be chosen to ensure a palpable muscle contraction and sensor tolerance. Each session will include a 2-minute warm-up and 2-minute cool-down of passive cycling. The unit automatically delivers enough stimulation to maintain a speed of 30 rotations per minute (rpm). Where this is not achieved, the leg cycle will assist the stimulated movement to maintain a speed of 30 rpm.
  Arms: Intervention

SUMMARY:
Spinal cord injury (SCI) is a devastating, life-altering injury; requiring tremendous changes in an individual's lifestyle. Cycling, provides an ideal way for individuals with SCI to exercise and address the long-term consequences of SCI by targeting the lower extremity muscles. Cycling with the addition of functional electrical stimulation (FES) allows persons with paralysis to exercise their paretic or paralysed leg muscles. The Queen Elizabeth National Spinal Injury Unit (QENSIU) in Glasgow offers FES cycling for people with spinal cord injuries, which combines functional electrical stimulation (FES) with a motorised ergometer that allows repetitive cycling activity. It stimulates muscles with electrodes attached to the skin, producing muscle contractions and patterned activity. So far no previous randomised control trials on FES cycling in the acute SCI population have reported changes in ability to undertake activities of daily living or the trunk balance.

DETAILED DESCRIPTION:
Up to 12 participants admitted to the QENSIU will be recruited to the study. They will be randomised to the intervention (n=8) or control group (n=4). The intervention group will receive 6 weeks FES cycling training in addition to usual care; the control group will receive usual care only. Outcome measures: Spinal Cord Injury Functional Ambulation Inventory, The Spinal Cord Independence Measure, ASIA Impairment Scale, Handheld dynamometry, 10-Metre Walking Test, Timed Up and Go Test, Trunk Impairment Scale, Modified Ashworth scale, Modified Tardieu Scale, the Patients Global Impression of Change.

ELIGIBILITY:
Inclusion Criteria:

* identified as being medically stable by the treating consultant,
* within the first 6 weeks post-injury,
* able to sit for 2 hours in a wheelchair,
* over 18 years old,
* acquired non progressive SCI - traumatic, spinal cord stroke, surgical injury,
* an incomplete SCI, graded as American Spinal Injury Association (ASIA) B (motor complete, sensation present below the lesion); C (some but not useful motor function) or D (useful motor function present),

Exclusion Criteria:

* acute condition impairing participant's ability to cycle (eg, leg fracture),
* proven or suspected neuromuscular weakness affecting the legs due to another condition (eg, stroke or Guillain-Barré syndrome),
* unable to follow instruction in English
* symptomatic cardiac disease,
* ventilator dependency,
* severe spasticity,
* uncontrolled autonomic dysreflexia,
* possible, suspected or confirmed pregnancy,
* likely to be discharged before the end of the exercise intervention.
* unable to tolerate the sensation of FES

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change in Spinal Cord Injury Functional Ambulation Inventory (SCI- FAI) | baseline, 6 weeks, 12 weeks
  It consists of three components: gait parameter, assistive device use and walking ability. The gait parameter component is scored out of 20, 10 points for each of the right and left sides. The assistive device component is scored out of 14 (7 points for each side), and assesses upper and lower extremities in addition to the left and right limbs. Scores within each component are summed. Component scores range from 0 to 20 in the gait parameter component, 0 to 14 in the assistive device component, and 0 to 5 in the walking mobility component. The SCI-FAI is a reliable, valid and sensitive measure of walking ability in individuals with spinal cord injury.

SECONDARY OUTCOMES:
The Spinal Cord Independence Measure (SCIM III) | baseline, 6 weeks, 12 weeks
  composed of 19 items that assesses 3 domains: self-care, respiration and sphincter management and mobility. The total SCIM scores range from 0 to 100.
ASIA Impairment Scale | baseline, 6 weeks, 12 weeks
  The ASIA impairment scale classifies motor and sensory impairment that results from a spinal cord injury. It divides spinal cord injuries into 5 categories: A-E. A- Complete - No motor or sensory function in the lowest sacral segment (S4-S5). B- Incomplete - Sensory function below neurologic level and in S4-S5, no motor function below neurologic level. C- Incomplete - Motor function is preserved below neurologic level and more than half of the key muscle groups below neurologic level have a muscle grade less than 3. D- Incomplete - Motor function is preserved below neurologic level and at least half of the key muscle groups below the neurologic level have a muscle grade >3. E- Normal - Sensory and motor function is normal
Handheld dynamometry (HDD) | baseline, 6 weeks, 12 weeks
  will be used to quantify the strength of the knee extensors, knee flexors, hip flexors, hip abductors, and ankle plantar flexors of both legs. The order of testing will be constant across testing sessions and position of patient and assessor standardised. Three trials will be performed on each muscle group. Prevention of muscle fatigue will be achieved by a 30-second recovery period after each trial and 2 minutes of rest between evaluations of the muscle groups. One or 2 trials will be used to familiarize the participants with the testing procedures before the actual strength measurements of each muscle group.
10-Metre Walking Test (10MWT) | baseline, 6 weeks, 12 weeks
  The total marked distance will be 14 meters and, to allow for acceleration and deceleration, participants will be timed over the middle 10 meters. Participants will walk the distance twice and the average of 2 trials will be measured. They will be asked to walk the distance as fast and safely as possible. The participant should perform this test with their assistive devices as appropriate.
Timed Up and Go (TUG) Test | baseline, 6 weeks, 12 weeks
  assesses mobility, balance, walking ability and falls risk. It measures, in seconds, the time taken by an individual to stand up from a standard arm chair (approximate seat height of 46 cm, arm height 65 cm), walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair, and sit down.
Trunk Impairment Scale (TIS) | baseline, 6 weeks, 12 weeks
  is a 17-item measure for assessing the level of motor impairment of the trunk e.g. coordination and sitting balance (static and dynamic). The scores range from 0 to 23 with lower scores indicating high levels of motor deficit in the trunk
Modified Ashworth scale (MAS) | baseline, 6 weeks, 12 weeks
  is a scale used to measure the level of spasticity in people with neurological conditions (ASHWORTH 1964). The MAS scores range from 0 to 4, with higher scores indicating an increase in muscle tone.
  0 No increase in muscle tone.
  1 Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension.
  1+ Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM.
  2 More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved.
  3 Considerable increase in muscle tone, passive movement difficult. 4 Affected part(s) rigid in flexion or extension
Modified Tardieu Scale (MTS) | baseline, 6 weeks, 12 weeks
  the MTS is a valid, reliable scale for measure the level of spasticity in patient with neurological conditions (Li, Wu, and Xiong 2014). Akpinar et al. (Akpinar et al. 2017) suggests its utility as a complementary tool when assessing spasticity in SCI patients. The MTS assesses the response of the muscle to different velocities of stretch in terms of quality and angle of the muscle tested. In terms of quality of muscle reaction, the score ranges from 0 to 5, where a score of 0 means that the muscle is not spastic while a score of 5 means that the muscle is spastic and immobile. In terms of angle of muscle reaction, the score is R1 or R2, where R1 means the joint demonstrates limited passive range of motion while R2 means the joint demonstrate full passive range of motion.
the Patients Global Impression of Change | 12 weeks
  PGIC is a 7-point, patient reported scale which evaluates all aspects of the patients' health and assesses if there has been an improvement or decline in clinical status. Patients rate their change as "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse" or "very much worse"

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Dybus, PhD, Principal Investigator — Glasgow Caledonian University
Locations (1):
- The Queen Elizabeth National Spinal Injuries Unit, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No